CLINICAL TRIAL: NCT05308927
Title: French Registry of Children Treated With Norditropin® for Short Stature Associated With Noonan Syndrome
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GH-4831; U1111-1264-1805 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-03-14; First posted 2022-04-04 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Noonan Syndrome
MeSH Terms: conditions — Noonan Syndrome | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Incident patients: Children initiated Norditropin® upon their inclusion in the study but independently from the decision to participate in this study
  Interventions: Drug: Norditropin
- Prevalent patients - finished growth upon inclusion: Children were already treated with Norditropin® before their inclusion in the study and finished their growth upon their inclusion. Data collected retrospectively from medical records
  Interventions: Drug: Norditropin
- Prevalent patients - not finished growth upon inclusion: Children were already treated with Norditropin® before their inclusion in the study and did not finish their growth upon inclusion. Data collected both retrospectively and prospectively
  Interventions: Drug: Norditropin

INTERVENTIONS:
Drug: Norditropin — Patients will be treated with commercially available Norditropin® according to routine clinical practice at the discretion of the treating physician.
  Other Names: Somatropin

SUMMARY:
This is a non-interventional registry of children treated with Norditropin® for short stature due to Noonan Syndrome (NS). This study aims to provide data on long-term growth evolution and safety of Norditropin® as well as Health Related Quality of Life (HRQoL) data. This registry will include the entirety of children treated with Norditropin® for short stature due to NS over the inclusion period. The decision to initiate treatment with commercially available Norditropin® is made by the patient/parents/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical and/or genetic diagnosis of NS
* Patients who are treated with Norditropin® (already treated or initiating) and who are followed in a participating center
* The decision to initiate treatment with commercially available Norditropin® has been made by the patient/parents/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study

Exclusion Criteria:

* Patients/Parents/LAR opposed to the collection and processing of their children's medical data
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The registry will include children treated with Norditropin® for short stature due to NS.
Sampling Method: Non-Probability Sample
Enrollment: 221 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2028-03-17 (Estimated); Study Completion 2028-03-17 (Estimated)

PRIMARY OUTCOMES:
Change in height standard deviation score | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in standard deviation scores (SDS) ranging from -10 to +10

SECONDARY OUTCOMES:
Number of adverse drug reactions (ADR) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Count of events
Number of serious adverse drug reactions (SADR) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Count of events
Number of serious adverse events (SAE) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Count of events
Number of adverse events (AE) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Count of events
Education | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Number of participants is measured under the categorical variables - standard education, education with assistance and educational measures
School level | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Number of participants is measured under the variables - preschool, elementary school, secondary school and high school
Educational measures | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Number of participants is measured under the categorical variables - physiotherapy, psychomotricity, occupational therapy and speech therapy
Tanner stage | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured as units on scale. 3 sub-scales used - Pubic hair scale, Female breast development scale and Male external genitalia scale. Tanner stages range from Stage 1 to 5 with Tanner Stage 1 corresponding to the pre-pubertal form and Tanner Stage 5 corresponding to the final adult form
Change in pulse rate | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in beats per minute
Change in diastolic blood pressure | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in millimeters of Mercury (mm Hg)
Change in systolic blood pressure | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in mm Hg
Change in corrected QT-interval (Electrocardiogram) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in millisecond (msec)
Change in echocardiogram parameters (mm) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Change in Left ventricular interventricular septal maximum thickness in diastole and Left ventricular end diastolic diameter is measured in millimeter (mm)
Change in echocardiogram parameters (%) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Change in Left Ventricular Fractional Shortening (LVFS) and Left Ventricular Ejection Fraction (LVEF) is measured in percentage (%)
Change in echocardiogram parameters (cm/s) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Change in Diastolic function (Ea and Aa) measured in centimeters per second (cm/s)
Change in complete blood count (CBC) (g/dL) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Change in Haemoglobin (Hb) measured in grams per deciLiter (g/dL)
Change in CBC (G/L) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Change in white blood cells, lymphocytes, monocytes and platelets measured in grams per liter (G/L)
Change in Insulin-like growth factor 1 (IGF-1) level (ng/ml) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in nanograms per milliliter (ng/ml)
Change in IGF-1 level (SDS) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in SDS
Change in Haemoglobin A1c (HbA1c) level | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in %
Change in fasting insulin level | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in milligrams per deciliter (mg/dL) or milli-international units per litre (mUI/L)
Change in fasting blood glucose level | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in mg/dL or g/L or millimoles per litre (mmol/L)
Change in fasting total cholesterol | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in mg/dl or g/L or mmol/L
Change in fasting triglycerides | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in mg/dL or g/L or mmol/L
Change in fasting high-density lipoproteins (HDL) cholesterol | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in mg/dL or g/L or mmol/L
Change in fasting low-density lipoproteins (LDL) cholesterol | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in mg/dL or g/L or mmol/L
Change in fasting total cholesterol/HDL ratio | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Ratio of fasting total cholesterol and HDL
Change in inhibin B | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in picograms per milliliter (pg/mL)
Change in Anti-Müllerian Hormone (AMH) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in milligrams per milliliter (mg/mL)
Change in Luteinizing Hormone (LH) (female from 8 years old and male from 9 years old) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in mg/mL
Change in Follicle-Stimulating Hormone (FSH) (female from 8 years old and male from 9 years old) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in International units per litre (UI/L) or mUI/mL
Change in oestradiol (female from 8 years old and male from 9 years old) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in pg/mL
Change in testosterone (female from 8 years old and male from 9 years old) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in ng/mL
Change in dose of Norditropin® treatment | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in milligram per kilogram per day (mg/kg/day)
Frequency of injections of Norditropin® treatment per week | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Count of events
Number of modifications (change in dosage/ temporary stop) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Count of events
Reasons for treatment modifications | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in number of participants under categorical variable - safety (occurrence of ARs or AEs), growth too fast, growth too slow, patient's or parents/LAR choice; and other
Duration of temporary stop | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in months
Total duration of Norditropin® treatment | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in years
Total cumulative dose of Norditropin® treatment | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in mg/kg
Type and number of concomitant treatments | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Count of events
Type and number of concomitant treatments linked to an adverse event | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Count of events
Change in weight | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in SDS
Change in body mass index (BMI) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in kilogram per square metre (kg/m^2)
Change in bone age | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in year
Change in height velocity (cm/year) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in cm/year
Change in height velocity (SDS/year) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Measured in SDS/year
Type and number of NS comorbidities | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  Number of participants measured under categorical variables - Cardiac defects including pulmonary valve stenosis and hypertrophic cardiomyopathy, Orthopaedic issues (pectus, scoliosis) and Anorchia in males
Change in Health-Related Quality of Life (HRQoL) score (PedsQL) | From start of Norditropin® treatment (day 0) until end of follow-up (up to 6 years)
  PedsQL score used to assess the HRQoL, ranges from 1 to 100 (higher scores indicate better HRQoL)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (3):
- France (3):
  - Centre Hospitalier Universitaire D'Angers-2, Angers
  - Ap-Hp-Hopital de Bicetre-2, Le Kremlin-Bicêtre
  - Hopital Des Enfants-2, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com